CLINICAL TRIAL: NCT02389049
Title: Research Genetic Testing for Primary Ciliary Dyskinesia Using a Panel of Genes
Brief Title: Genetics of Primary Ciliary Dyskinesia
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-1225; U54HL096458-11 (NIH)
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Primary Ciliary Dyskinesia; Kartagener Syndrome
Keywords: Primary Ciliary Dyskinesia; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood or buccal samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is designed to study DNA sequencings for mutations in a research genetic test panel of genes (which contains all 32 known and/or published genes associated with PCD). The study aims to show that about 70% of PCD patients have biallelic mutations in one of these genes. This project will enroll patients who have already had a clinical evaluation, and have clinical features consistent with PCD.

DETAILED DESCRIPTION:
The investigators have established a Consortium of 9 geographically-dispersed clinical research sites to study rare disease of the airways, including Primary Ciliary Dyskinesia (PCD). PCD is a genetic disorder with defective mucociliary clearance (MCC), sinus and pulmonary disease with chronic infection, and organs located on the wrong side of the body in about 50% of patients (Kartagener Syndrome). Lung disease occurs early in children with PCD, but establishing a diagnosis remains a major challenge, based on the traditional approaches of using electron microscopy and/or ciliary waveform analysis to define abnormalities of ciliary ultrastructure and/or function.

For this study, blood or buccal samples for DNA will be collected and genetic testing in patients with known or suspected PCD will be performed. This study can include term neonates with respiratory distress of unknown etiology and features of PCD, particular laterality defects (situs inversus or heterotaxy). The key hypothesis for this study is that a genetic test panel of 32 genes will confirm a diagnosis in most patients with PCD.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has ≥ 2 clinical features (+/- lab) characteristic of PCD, including:

  * Neonatal respiratory distress after term (or near-term) birth
  * and/or laterality defect ( situs inversus or heterotaxy)
  * and/or daily wet cough before 6 months of age
  * and/or middle ear disease
  * and/or chronic nasal congestion before 6 months of age
  * and/or bronchiectasis
  * and/or male infertility due to sperm tail dysfunction
  * and/or low nasal nitric oxide levels (<77 nanoliters/minute)
  * and/or defective ciliary ultrastructure

Exclusion Criteria:

* Known diagnosis of cystic fibrosis with classic clinical presentation and elevated sweat chloride levels and/or two known disease-causing Cystic Fibrosis transmembrane conductance regulator (CFTR) mutations, or documented primary or acquired immunodeficiency.
* Known explanation for bronchiectasis (and other clinical features), such as α1-antitrypsin deficiency (ZZ or ZS), inflammatory bowel disease or rheumatoid arthritis.
* Any patient who is unwilling or unable to provide consent or to comply with the testing required in this protocol

A participant should not be in the study if they have not had a standard clinical evaluation to address other potential causes of chronic oto-sino- pulmonary disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants should have 2 or more clinical features of PCD.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2015-02; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Confirm PCD diagnosis in patients using a panel of 32 genes | Up to 5 years
  The primary objective is to perform research genetic (Ampliseq panel) testing in patients who are known or suspected to have PCD, based on previous research or future clinical and lab characterization by certified clinical research sites. We will define the prevalence of biallelic PCD-causing mutations in patients who fulfill criteria of very high likelihood of PCD, as well as prevalence in other patients with some features of PCD. We anticipate successful completion of this objective will provide the foundation for development of clinically available genetic test panels, particularly as additional PCD genes are identified.

SECONDARY OUTCOMES:
Identify patients with PCD who do not have a biallelic PCD-causing mutation | Up to 5 years
  The secondary objective is to perform research genetic testing to identify patients with PCD who do not have biallelic PCD-causing mutations in known PCD genes, so they can be exome sequenced to discover novel genes associated with PCD. We anticipate that successful completion of this objective will enable the development of more extensive genetic test panels that are more robust to diagnose PCD.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knowles, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (8):
- United States (6):
  - Stanford University, Palo Alto, California
  - The Children's Hospital, Denver, Aurora, Colorado
  - Riley Hospital for Children, Indianapolis, Indiana
  - Washington University, St. Louis, St Louis, Missouri
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital and Regional Medical Center, Seattle, Seattle, Washington
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Kaspy KR, Dell SD, Davis SD, Ferkol TW, Rosenfeld M, Sagel SD, Milla C, Olivier KN, Barber AT, Wee W, Lin FC, Li L, Rampakakis E, Zariwala MA, Knowles MR, Leigh MW, Shapiro AJ. Situs Ambiguus Is Associated With Adverse Clinical Outcomes in Children With Primary Ciliary Dyskinesia. Chest. 2024 May;165(5):1070-1081. doi: 10.1016/j.chest.2023.12.005. Epub 2023 Dec 9. PMID 38072392